CLINICAL TRIAL: NCT05568745
Title: Balloon + Oxytocin Versus Oral Misoprostol to Induce Labor in Case of Premature Rupture of Membranes (PROM) at Term in Nulliparous: a Randomized Controlled Trial (RUBAPRO2).
Brief Title: Balloon + Oxytocin Versus Oral Misoprostol to Induce Labor in Case of PROM (RUBAPRO2)
Acronym: RUBAPRO2
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PHRC N 2020 GALLOT; 2022-A01479-34 (Other: ANSM); 2022-501142-30-00 (Other: UECT - ANSM)
Record Dates: First submitted 2022-09-26; First posted 2022-10-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Induction of Labor; Cervical Ripening; Premature Rupture of Fetal Membranes; Nulliparous
Keywords: premature rupture of membranes; labour induction; unfavourable cervix; cervical ripening balloon; pharmacological cervical ripening; misoprostol
MeSH Terms: conditions — Fetal Membranes, Premature Rupture | interventions — Oxytocin; Misoprostol

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, controlled, open-label therapeutic trial with two parallel arms.
Masking Description: Masking is impossible because of the nature of the device studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balloon+oxytocin (Experimental): Mecanical cervical ripening will be done by transcervical balloon (Teleflex French Dufour catheter CH20 reference 174000). Oxytocin will be started 6 hours after balloon insertion. At H12 balloon will be removed and induction continued by oxytocin alone.
  Interventions: Device: Balloon for cervical ripening (Teleflex French Dufour catheter CH20 reference 174000); Drug: Oxytocin
- Oral misoprostol (Active Comparator): Patients will receive misoprostol 25 micrograms given orally (oral prostaglandin E1). The same dose will be given every 2 hours until beginning of labor with a maximum of 8 administrations. (Oxytocin can be started at least 4 hours after the last misoprostol administration if patient remains not in labour.)
  Interventions: Drug: Misoprostol Oral Tablet

INTERVENTIONS:
Device: Balloon for cervical ripening (Teleflex French Dufour catheter CH20 reference 174000) — Balloon catheter is inserted by a resident or a physician under visual control. The expected volume injected in the balloon probe is 60 mL. No traction is performed on the catheter. The catheter is left in place for a maximum of 12 hours.
  Arms: Balloon+oxytocin
Drug: Oxytocin — Intravenous oxytocin addition (preceded or followed by epidural analgesia on patient's request) will be performed 6 hours after insertion of balloon catheter. Oxytocin is administered as an intravenous infusion (5 IU of oxytocin in 49 mL of 5% glucose*) at the lowest possible dose with the aim of achieving a maximum of three to four contractions per ten minutes. After appropriate uterine activity has been achieved, the rate of the oxytocin infusion is decreased or stopped.
  Arms: Balloon+oxytocin
Drug: Misoprostol Oral Tablet — Patients will receive misoprostol 25 micrograms given orally (oral prostaglandin E1). The same dose will be given every 2 hours until beginning of labor with a maximum of 8 administrations.
  Arms: Oral misoprostol

SUMMARY:
Premature rupture of membranes (PROM) at term complicates 6 to 22% of singleton pregnancies. Spontaneous labour occurs in 60-67% of these patients within 24h. If no effective uterine contraction occurs, induction of labour (IOL) is the strategy recommended by the French as well as the American College of Obstetricians and Gynecologists. The optimal strategy for IOL in case of PROM with an unfavourable cervix remains unknown and none of the studies conducted in nulliparous women showed the superiority of one induction method over another.

In the current project, we aimed to determine (1) if IOL with association of balloon catheter and oxytocin after 6 hours could increase the rate of delivery < 24h versus low dose of oral misoprostol (25 µg oral PGE1 every 2h) in case of PROM at term in nulliparous women and (2) patient satisfaction using EXIT survey assessed before hospital discharge.

DETAILED DESCRIPTION:
Context : Premature rupture of membranes (PROM) at term complicates 6 to 22% of singleton pregnancies. Spontaneous labour occurs in 60-67% of these patients within 24hours. If no effective uterine contraction occurs, induction of labour (IOL) is the strategy recommended by the French as well as the American College of Obstetricians and Gynecologists. The optimal strategy for IOL in case of PROM with an unfavourable cervix remains unknown and none of the studies conducted in nulliparous women showed the superiority of one induction method over another1. Oral misoprostol (ProstaglandinE1, PGE1) usually demonstrated the lowest rate of c-section after IOL in general population and balloon catheter was associated with the lowest rate of uterine hyperstimulation. Recently, a comparison 1 to 1 between these two methods was conducted in singletons with comparable results. Despite recent studies demonstrating no higher risk of infectious complications using mechanical device in the context of PROM, only prostaglandins and oxytocin are usually recommended. Recently, Devillard et al. demonstrated that the combination of balloon catheter plus oxytocin systematically infused after 6 hours increased the rate of delivery <24h compared to dinoprostone vaginal insert group (90% versus 57.5% respectively) and decreased the time between induction and delivery in nulliparous group (17.0hours versus 26.5hours).

In the current project, we aimed to determine (1) if IOL with association of balloon catheter and oxytocin after 6 hours could increase the rate of delivery < 24hours versus low dose of oral misoprostol (25 µg oral PGE1 every 2h) in case of PROM at term in nulliparous women and (2) patient satisfaction using EXIT (EXperience of Induction Tool) survey assessed before hospital discharge.

We hypothesized that the rate of delivery < 24hours will be 15% higher in the group induced with balloon + oxytocin (estimated around 85 %) compared to the misoprostol group (estimated around 70 %). Patient satisfaction concerning experience of IOL will be assessed using a validated survey- the EXperience of Induction Tool (EXIT) - translated in French language (Beckman et al., 2017). We aimed to demonstrate a difference greater than an effect-size of 0.25.

Objectives: The main objective is to demonstrate higher rate of vaginal birth <24hours by insertion of a balloon catheter + oxytocin after 6hours, versus low dose of oral misoprostol (25 µg oral PGE1 every 2hours) in case of unfavorable cervix beyond 12 hours of PROM in nulliparous and to compare patient satisfaction using EXIT survey translated in French language before hospital discharge.

The secondary objectives are:

* To compare the rate of caesarean sections in the two groups.
* To compare the safety related to women of both induction methods in terms of maternal morbidities, uterine hyperstimulation, maternal infections and other reported adverse events (AEs).
* To compare the safety related to neonates of both induction methods in terms of neonatal morbidities, neonatal infections and other reported AEs.

Study type: Multi-center, randomized, controlled, open-label therapeutic trial with two parallel arms.

Number of centers: 5

Study Description:

The study group is the balloon catheter group with addition of oxytocin as early as 6h after the catheter insertion. After 12 hours of balloon insertion, induction of labour is continued by oxytocin alone. The control group corresponds to induction with misoprostol 25µg given orally (oral prostaglandin E1). The same dose is delivered every 2 hours until labour onset with a maximum of 8 administrations. Oxytocin can be started at least 4 hours after the last misoprostol administration.

Patients will be assigned by random allocation on a 1:1 basis in permuted blocks to either treatment group or control group using a dedicated, password-protected, SSL-encrypted website. To minimize the risk of imbalance between the study groups, the randomization will be stratified by trial site.

Primary endpoint: Hierarchical primary endpoint: (1) Proportion of patients vaginally delivered <24h and (2) patient satisfaction using EXIT survey assessed before hospital discharge.

Number of patients: 520

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old,
* Pregnant, Gestational age ≥ 37 weeks
* Singleton pregnancy with cephalic presentation
* Nulliparous
* PROM without labour beyond 12 hours
* Unfavourable cervix (Bischop score < 6)
* Able to give her informed consent
* Ability to comply with the requirement of the study
* Covered by the French Social Security welfare system

Exclusion Criteria:

* Unable to understand French language
* Contraindication for vaginal delivery
* Loss of meconium amniotic fluid (LA)
* Temperature > 38.2°C
* Intrauterine infection
* IUGR with Doppler anomaly
* Fetus with expected polymalformative syndrome
* Scarred womb
* Suspicion of genital herpes
* Known HIV seropositivity
* Placenta praevia
* Fetal death
* Abnormal FHR (Fetal Heart Rate)
* Contraindication to misoprostol:

  * Allergy or hypersensibility
  * Suspicion or confirmation of a scarred uterus following past surgical intervention
  * Renal insufficiency
  * Malformation of the uterus
* Contraindication to balloon:

  * Vasa praevia, placenta praevia
  * Invasive cervical cancer
* Contraindication to oxytocin

  * Allergy or hypersensibility
  * Dystocia
  * Fragility or excessive distension of the uterus
  * Uterine hypertonia or fetal distress when delivery is not imminent
  * Cardiovascular disorders and severe preeclampsia
  * Predisposition to amniotic embolism (in utero fetal demise, abruption).
* Patient subject to a legal protection order (curatorship or tutorship)
* Refusal to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Vaginal delivery <24hours | at birth
  Proportion of patients vaginally delivered <24hours (in %)
Patient satisfaction | up to 4 days
  Satisfaction of women concerning method of induction by the EXperience of Induction Tool (EXIT) validated in french language.

SECONDARY OUTCOMES:
Duration from rupture to beginning of induction | at birth
  in hours
Duration between IOL and delivery | at birth
  in hours
Duration of balloon exposure or misoprostol exposure | at birth
  in hours
Misoprostol received | at birth
  Total dose of misoprostol received (in µg)
Bishop score on balloon removal | at birth
  (comprised between 0 and 13)
Balloon in place (yes/no) | at birth
  Rate of balloon in place (%) at 12 hours after the beginning of induction
Duration between induction and full cervical dilatation | at birth
  Duration (in hours)
Mode of delivery | at birth
  Rate in %
Post-partum hemorrhage | up to 4 days
  Rate in %
Rate of fever | during labor
  Rate in %
Rate of patients experiencing episode(s) of uterine hyperstimulation | during labor
  Rate of patients experiencing episode(s) of uterine hyperstimulation (%) during labour (defined by the necessity to interrupt oxytocin and/or to inject pharmacological agents in the context of excessive number of contractions with or without abnormal FHR),
Endometritis | up to 4 days
  Rate of endometritis in %
Duration of hospital stay | up to 4 days
  Duration (in days)
Birth weight of the newborn | at birth
  in grammes
Apgar score < 7 | 5min after birth
  Neonatal endpoint (yes/no)
pH umbilical artery | at birth
  pH at the umbilical artery
Base defect and lactate (umbilical artery) | at birth
  mmol/L
Neonatal tranfer | up to 4 days
  Rate of neonatal transfer to intensive care unit or neonatology unit
maternal-fetal infection | up to 4 days
  Rate of maternal-fetal infection in %

CONTACTS AND LOCATIONS:
Overall Officials: Denis Gallot, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (5):
- France (5):
  - CHU de Bordeaux, Bordeaux
  - CHU de Clermont-Ferrand, Clermont-Ferrand
  - Assistance Publique Hôpitaux de Paris- CHU Bicêtre, Le Kremlin-Bicêtre
  - CHU de Saint Etienne, Saint-Etienne
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Derived] Rouzaire M, Triolaire A, Vayssiere C, Sentilhes L, Barjat T, Luton D; Groupe de Recherche en Obstetrique et Gynecologie (GROG) Investigators; Davoust E, Cabrespine A, Pereira B, Gallot D. Balloon plus oxytocin or oral misoprostol for labour induction in prelabour rupture of membranes (PROM): protocol for a randomised controlled trial (RUBAPRO2). BMJ Open. 2026 Jan 27;16(1):e110425. doi: 10.1136/bmjopen-2025-110425. PMID 41592839